CLINICAL TRIAL: NCT01786967
Title: Understanding the Response to Fesoterodine Through Genetic Evaluation in the Elderly
Brief Title: Understanding the Response to Fesoterodine Through Genetic Evaluation in the Elderly (URGE)
Acronym: URGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-2066; 1R03AG042335-01 (NIH); Pro00036147 (Other: UNC)
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2018-12

CONDITIONS: Urge Urinary Incontinence
Keywords: overactive bladder; urge urinary incontinence; pharmacogenetics
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fesoterodine Fumarate (Experimental): Participants will receive 4 mg of study drug for first 2 weeks, and then 8 mg of study drugs for 2 weeks.
  Interventions: Drug: Fesoterodine Fumarate

INTERVENTIONS:
Drug: Fesoterodine Fumarate — FDA approved anticholinergic medication used for treatment of urge urinary incontinence
  Other Names: Toviaz

SUMMARY:
Urge urinary incontinence, characterized by unpredictable and embarrassing large volume urine leakage, is a major health issue for elderly women, as it is incredibly common and significantly impairs quality of life. Although anticholinergic medications are the most common therapy, the investigators are unable to predict an individual's response to a particular drug in terms of both effectiveness and side effects. Through genetic evaluation, the investigators have the potential to personalize and optimize drug therapy for millions of elderly women suffering from urge incontinence.

DETAILED DESCRIPTION:
Urge urinary incontinence (UUI), characterized by unpredictable and embarrassing large volume urine leakage, is a major public health burden to elderly women, given its high prevalence, impairment of quality of life, associated caregiver burden, and substantial economic costs. UUI is significantly more prevalent in older adults and disproportionately affects women, with a prevalence of 19% in community-dwelling women over 65 and 60-78% in long-term care female residents.

Anticholinergic medications are the most common first-line therapy for UUI. Although numerous trials have demonstrated that anticholinergics are efficacious for UUI, the response to these medications is variable, as their effectiveness is often limited by poor response or adverse events (AEs), such as cognitive impairment or constipation, which are particularly problematic in older adults. Furthermore, a comprehensive systematic review concluded that no one drug is definitively superior, leaving clinicians without any evidence to guide decision-making regarding drug choice. As a result, UUI pharmacotherapy is empiric and not personalized, even though it is clear that individual variations exist in both response and toxicity. The treatment of UUI is especially challenging in the geriatric population, given their higher risk for AEs, polypharmacy, and pharmacokinetic changes that occur with age. The ability to predict which elderly women with UUI will experience low efficacy or develop significant adverse events from anticholinergic medications would be a paradigm shift in the therapeutic practice to this highly prevalent and bothersome condition.

Pharmacogenetics may provide insight into how to predict response to anticholinergic UUI therapy. Research has already shown that genetic differences in drug metabolism impact a patient's drug response. For example, "fast metabolizers" may metabolize the drug so rapidly that therapeutic levels are never reached, limiting effectiveness. In contrast, "slow metabolizers" may develop high drug concentrations, resulting in significantly more AEs. While pharmacogenetic research exists for numerous classes of drugs, including anticoagulants, selective serotonin-reuptake inhibitors,14 beta-blockers, immunosuppressants and opioids, this type of translational research does not exist for anticholinergics for UUI. Thus, this proposed project represents a novel concept and unique opportunity to dramatically change UUI pharmacotherapy.

Fesoterodine is an ideal anticholinergic medication to launch a pharmacogenetic study in this field. Fesoterodine's active metabolite, 5-hydroxymethyl tolterodine (5-HMT), is metabolized by a well-characterized cytochrome P450 (CYP) enzyme, CYP2D6. The CYP2D6 gene has several genetic variants, which result in different metabolizer statuses ranging from poor metabolizers (PM), intermediate metabolizers (IM), extensive metabolizers (EM), to ultrarapid metabolizers (UM). These different CYP2D6 profiles may be clinically important, as they may contribute to the variability in efficacy and AEs. In fact, pharmaceutical company data for fesoterodine demonstrated that PMs have a two-fold higher plasma concentration than EMs; however, no published data exist on how CYP2D6 metabolizer status correlates with clinical outcomes such as efficacy or AEs. The ability to use CYP2D6 metabolizer status to predict which individuals will experience low efficacy or develop AEs to fesoterodine, and to utilize alternative therapies in these women, would challenge existing therapeutic paradigms and would significantly advance clinical practice via a pharmacogenetic approach.

Specific Aim 1: To explore whether CYP2D6 metabolizer status can predict efficacy during 4 weeks of fesoterodine fumarate therapy in elderly women with UUI. All subjects will be started on fesoterodine 4mg for 2 weeks followed by 8mg for 2 weeks. The primary outcome will be patient-reported treatment response based on a 4-point scale utilized in phase III clinical trials.8,9 We hypothesize that women who rapidly metabolize fesoterodine based on CYP2D6 metabolizer status are more likely to have low efficacy.

Specific Aim 2: To explore whether CYP2D6 metabolizer status can predict moderate to severe adverse events during 4 weeks of fesoterodine fumarate therapy in elderly women with UUI. In the same study design as Aim #1, we will identify subjects with moderate to severe fesoterodine-related AEs. We hypothesize that women who are CYP2D6 poor metabolizers are more likely to have moderate to severe AEs.

Specific Aim 3: To utilize preliminary data from this pilot, proof-of-concept study to plan a future large-scale trial to predict outcomes of anticholinergic UUI therapy based on CYP2D6 metabolizer status. Data regarding efficacy rates, risk of moderate-severe AEs, and the impact of CYP2D6 metabolizer status on efficacy and AEs, in addition to information regarding recruitment, drop-out, and questionnaire burden, will critically inform the study design, outcome measures and sample size of future, definitive trials.

This proposal represents an innovative approach to pharmacotherapy for UUI, a highly prevalent condition with significant morbidity. Pharmacogenetics has tremendous potential to identify ideal candidates for anticholinergic UUI therapy and to distinguish individuals who may benefit from alternative treatment options. This pioneering pharmacogenetic research has the potential to lay the necessary groundwork for future long-term research which would optimize and personalize UUI therapy for millions of elderly women.

Design & Procedures:

Patient Population: All women aged 50 years or older who desire treatment for bothersome UUI will be approached for enrollment. Women with ≥ 3 UUI episodes on a 3-day voiding diary will be included. Although women who have previously failed fesoterodine will be excluded, those who have failed other UUI anticholinergics remain eligible after a 2-week washout period.

Subjects with auditory or visual sensory impairment will be included. If visual impairment exists, the research coordinator will provide assistance to complete the necessary documents. However, those who are unable to complete the study-related items and visits, such as women with cognitive impairment, based on the Mini-Cog validated questionnaire will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 50 years
* ≥ 3 UUI episodes on a 3-day voiding diary
* Urge-predominant incontinence, >50% of total incontinence episodes
* No history of failure to fesoterodine
* 2-week washout period if currently on an anticholinergic for UUI
* Willingness to avoid off-protocol UUI therapy during the study period
* Post Void Residual (PVR) <150 mL

Exclusion Criteria:

* Contraindications to fesoterodine (e.g., bladder outlet obstruction, narrow angle glaucoma, myasthenia gravis, severe hepatic or renal impairment)
* Inability to complete study-related items and visits - i.e., cognitive impairment based on Mini-Cog test score (exclude if score of 0 or 1-2 (Abnormal))
* Urinary retention requiring catheterization
* Symptomatic, untreated urinary tract infection not resolved prior to starting fesoterodine
* Botulinum toxin injection for UUI in the last year
* Current therapy with peripheral or sacral neuromodulation
* Neurologic conditions that may affect urinary function (stroke, multiple sclerosis, spinal cord injury, Parkinson's disease)
* Women taking potent CYP3A4 inhibitors

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Wu, MD, Principal Investigator — UNC-CH
Locations (1):
- UNC-Chapel Hill, Dept of Ob/Gyn, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fesoterodine Fumarate
Started | 61
Extensive Metabolizers | 54
Poor Metabolizers | 4
Metabolizer Status Undetermined | 3
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The number of participants who received the intervention
Groups:
- Fesoterodine Fumarate: Women aged 50 and older received 4mg of fesoterodine fumarate for 2 weeks followed by 8mg fesoterodine for 2 weeks.
Arm/Group | Fesoterodine Fumarate
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Functional Comorbidity Index Score [Median (Inter-Quartile Range); unit: units on a scale] — The Functional Comorbidity Index (FCI) consists of 18 diagnoses associated with diminishing function where 1 point is assigned for the presence of each diagnosis. Points are summarized for an overall score ranging from 0 to 18. Higher scores reflect the presence of a greater number of comorbid conditions.
  units on a scale | 3 [2.5 to 4.5]
Current smoker [Count of Participants; unit: Participants]
  Current smoker-Yes | 2
  Current smoker-No | 59
Katz ADL (Activities of Daily Living) score (total) [Median (Inter-Quartile Range); unit: units on a scale] — The Katz Index of Independence in Activities of Daily Living (Katz ADL) assesses functional status as a measurement of the client's ability to perform activities of daily living independently. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Participants are scored No or Yes (no=0 and yes=1) for independence in each of the six functions; thus, total scores range from 0 to 6, with a higher score indicating better function.
  units on a scale | 5 [5 to 5]
Lawton IADL (Instrumental Activities of Daily Living Scale) score (total) [Median (Inter-Quartile Range); unit: units on a scale] — The Lawton Instrumental Activities of Daily Living Scale (IADL) assesses skills that are more complex than the basic activities of daily living (ie Katz ADLs). There are 8 domains of function including telephone use, food preparation, housekeeping, laundering, transportation, responsibility for own medications and handling finances. Scores for each of the 8 domains range from 0 to 1 such that total scores range from 0 to 8, with higher scores indicating higher function.
  units on a scale | 8 [8 to 8]
Overactive bladder questionnaire - symptom bother [Mean (Standard Deviation); unit: units on a scale] — Overactive bladder questionnaire (OABq) short form is a validated questionnaire that assesses symptom bother from OAB as well as health-related quality of life impact from overactive bladder (condition of urinary urgency, frequency and/or urgency incontinence). Higher scores indicate greater symptom severity. Transformed scores range from 0-100.
  units on a scale | 68.1 (19.9)
Overactive bladder questionnaire - quality of life [Mean (Standard Deviation); unit: units on a scale] — Overactive bladder questionnaire (OABq) short form is a validated questionnaire that assesses symptom bother from OAB as well as health-related quality of life impact from overactive bladder (condition of urinary urgency, frequency and/or urgency incontinence). Subscales include coping, sleep and social. Higher scores indicate better health-related quality of life. Transformed scores range from 0-100.
  units on a scale | 48.0 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage With Treatment Success
Description: Treatment Success (Yes/No) was defined by the Treatment Benefit Scale (TBS). TBS is a 4-point scale which was dichotomized into Yes/No for the Treatment Success outcome. The scale asks participants to rate "My condition has been improved: 1= greatly improved, 2=improved, 3=not changed, 4= worsened." If a participant responded 1 (greatly improved) or 2 (improved), they were considered as a "Yes" for Treatment Success. If a participant responded 3 (not changed) or 4 (worsened), then they were considered as a "No" for Treatment Success.
Time Frame: 4 weeks
Population: Extensive and poor metabolizers are the two cohorts being compared. These cohorts were determined based on their CYP2D6 sequence. Only 58 subjects have data as 3 participants' sequencing did not yield a definitive metabolizer status.
Measure: Number; unit: percentage of participants
Groups:
- Extensive Metabolizers: Extensive metabolizer status was based on CYP2D6 sequence
- Poor Metabolizers: Poor metabolizer status was based on CYP2D6 sequence
Arm/Group | Extensive Metabolizers | Poor Metabolizers
Number analyzed (Participants) | 54 | 4
percentage of participants | 74.1 | 75.0
Statistical Analysis 1: Comparison: Extensive Metabolizers vs Poor Metabolizers; Null hypothesis was that there will be no difference in treatment benefit scale between the two groups; Test type: Superiority — This was a pilot study to provide preliminary data to inform future sample size estimates for a larger more definitive trial; p = 1.0, Fisher Exact; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.53 to 1.71]

2. Secondary Outcome: Percentage With Moderate to Severe Anticipated Drug Associated Adverse Events
Description: Outcome was defined as moderate to severe anticipated adverse events (AE) based on the NCI Common Terminology Criteria for Adverse Events (CTCAE). Each AE is graded 1-5 with Grade 1=mild AE, Grade 2=moderate AE, Grade 3=severe AE, Grade 4=life-threatening or disabling AE, grade 5=Death-related to AE. Any side effect grade >= 2 considered a moderate to severe AE. Anticipated AEs included dizziness, somnolence, insomnia, confusion, cognitive impairment, dry eyes, blurry vision, dry mouth, constipation, nausea, dyspepsia and urinary retention. Example: dry mouth grades per CTCAE: Grade 1=symptomatic without significant dietary alteration; unstimulated saliva flow > 0.2 mL/min; Grade 2=symptomatic and significant oral intake alteration; unstimulated saliva flow 0.1 to 0.2 mL/min; Grade 3=symptoms leading to inability to adequately aliment orally; IV fluids, tube feedings or total parenteral nutrition indicated; unstimulated saliva < 0.1 mL/min.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Extensive Metabolizers: Extensive metabolizer status is based on CYP2D6 sequence
- Poor Metabolizers: Poor metabolizer status is based on CYP2D6 sequence
Arm/Group | Extensive Metabolizers | Poor Metabolizers
Number analyzed (Participants) | 54 | 4
percentage of participants | 14.8 | 0.0
Statistical Analysis 1: Comparison: Extensive Metabolizers vs Poor Metabolizers; Null hypothesis was that there was no difference in the rate of moderate to severe adverse events; Test type: Superiority; p = 1.0, Fisher Exact; Risk Ratio (RR) = 0.85, 95% CI 2-sided [.76 to .95]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Metabolizer Status Undetermined: Metabolizer status was not able to be determined
Arm/Group | Extensive Metabolizers | Poor Metabolizers | Metabolizer Status Undetermined
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 5/54 | 0/4 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extensive Metabolizers (N=54) | Poor Metabolizers (N=4) | Metabolizer Status Undetermined (N=3)
Anticholinergic adverse events (Eye disorders) | 5 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a pilot study. Given the smaller size of the study population in this pilot trial, the number of poor metabolizers is low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT01786967/Prot_SAP_000.pdf